CLINICAL TRIAL: NCT02263339
Title: Aerobic Exercise to Improve Brain Metabolism in MS
Brief Title: Exercise & Brain Health in MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Rebecca Spain, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 10599
Record Dates: First submitted 2014-10-02; First posted 2014-10-13 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Multiple Sclerosis
Keywords: Exercise; MRI
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aerobic Exercise (Experimental)
  Interventions: Behavioral: Aerobic Exercise
- Stretching Program (Active Comparator)
  Interventions: Behavioral: Stretching
- Aerobic Exercise, Healthy Subjects (Active Comparator)
  Interventions: Behavioral: Aerobic Exercise- Healthy Subjects

INTERVENTIONS:
Behavioral: Aerobic Exercise — Each subject will exercise 30 minutes per session, four times per week for 8 weeks at the OHSU Human Performance Laboratory (HPL). Choice of treadmill or cycle ergometer for each subject will be made based on subject ability by the HPL staff and maintained for the duration of the study. Exercise intensity will be determined by training heart rate to be provided to the subject based on the anaerobic threshold during initial stress test. Throughout the study, patients will be instructed not to alter their diet or baseline level of activity.
  Arms: Aerobic Exercise
Behavioral: Stretching — Each subject will follow a self-guided stretching program 30 minutes per session, four times per week for 8 weeks. The initial session will be supervised at the OHSU Human Performance Laboratory (HPL) and additional supervised sessions will occur every 2 weeks to support compliance with the program. Throughout the study patients will be instructed not to alter their diet or baseline level of activity.
  Arms: Stretching Program
Behavioral: Aerobic Exercise- Healthy Subjects — Each subject will follow a self-guided aerobic exercise program 30 minutes per session, four times per week for 8 weeks. The initial session will be supervised at the OHSU Human Performance Laboratory (HPL) and additional supervised sessions will occur every 2 weeks to support compliance with the program. Throughout the study patients will be instructed not to alter their diet or baseline level of activity.
  Arms: Aerobic Exercise, Healthy Subjects

SUMMARY:
The purpose of this study is to learn more about multiple sclerosis (MS). The investigators are studying whether aerobic exercise is better than a stretching program at improving brain health in people with MS. We want to learn:

1. If it is safe and practical for people with MS to participate in an aerobic exercise program with the goal of increasing cardiac fitness. Cardiac fitness is measured with exercise stress tests at the beginning and end of the study.
2. If aerobic exercise improves brain metabolism, a reflection of brain health, more than stretching. Brain metabolism is measured by MRIs at the beginning and end of the study.

There is a 50% chance of being in the aerobic exercise or the stretching program.

There are between 8 and 36 visits to OHSU, depending on the intervention group. The total duration of the study is at most 21 weeks.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a disease of brain, spinal cord and optic nerves. Current MS therapies reduce the frequency and severity of MS flare-ups, but do not help MS in later stages of disease characterized by slow progression of disability. One obstacle to developing therapies for progressive aspects of disease is a lack of ability to measure progression and brain repair.

A new MRI technique developed by Bill Rooney, PhD, (co-investigator, OHSU Advanced Imaging Resource Center) looks at brain health by measuring levels of phosphorous. Phosphorous levels are thought to reflect energy stores produced by brain cells. The healthier the brain, the greater the energy stores seen as higher the levels of phosphorous on imaging. Dr. Rooney has shown decreased levels of phosphorous on brain MRIs from people with MS. We propose that therapies that boost brain cell health will lead to an increase in brain cell energy stores and be reflected by an increase in phosphorous levels on MRI spectroscopy.

In order to test whether improvements in brain energy stores can be seen as increased phosphorous levels, we will use a therapy known to improve energy stores in muscles and see if it also does so in the brain. We measure how much aerobic exercise increases energy stores in muscles by measuring oxygen utilization during an exercise stress test. Therefore in this study, we will see if the aerobic exercise that improves muscle energy stores (seen as an increase in oxygen utilization) corresponds to an increase in brain energy stores (seen as an increase in phosphorous levels).

Specific Aim 1. To determine if it is safe and feasible to conduct an aerobic exercise intervention in MS patients to achieve an increase in oxygen utilization by 5-15%.

Hypothesis: An MS cohort undergoing a structured aerobic exercise program will increase their aerobic capacity by 5-15% as measured by oxygen utilization testing and not experience adverse events related to the exercise program.

Specific Aim 2. To determine if brain phosphorous levels by MR spectroscopy before and after an aerobic exercise intervention increases in association with increases in oxygen utilization.

Hypothesis: Aerobic exercise will increase energy stores in both muscles and the brain. Body energy stores will be measured by oxygen utilization testing and brain energy stores by phosphorous levels. We expect that increases in by oxygen utilization after a structured exercise program will be associated with increases in phosphorous levels. We do not expect increases in either by oxygen utilization or phosphorous levels in an MS cohort matched for sex and baseline aerobic capacity that participates in a non-aerobic stretching program of the same duration and intensity.

Outcome measures: The primary outcome is change in brain phosphorous levels by MRI spectroscopy. The secondary outcomes are changes in oxygen utilization levels, walking and balance tests, and changes in cognitive function and energy levels.

Methods: Participants will be enrolled over a 1 year period. Potential subjects will undergo a baseline exercise stress test for oxygen utilization. Participants matched by sex and baseline oxygen utilization level will undergo a baseline MRI spectroscopy study and then be randomly assigned to either an aerobic exercise program or a self-guided stretching program. The aerobic exercise program consists of supervised 30 minute sessions of either treadmill or stationary bicycle exercise, 4 days per week for 8 weeks. The self-guided home stretching program consists of 30 minute sessions, 4 days a week for 8 weeks with supervised sessions occurring every 2 weeks. All participants will undergo a final exercise stress test and MRI spectroscopy. Only participants who are matched and assigned to either exercise or stretching groups will undergo MRI testing and receive payment for participation.

ELIGIBILITY:
Inclusion Criteria:

i. Physician-confirmed diagnosis of relapsing-remitting MS ii. > 18 years old iii. Expanded Disability Status Scale (EDSS) < 4.0 iv. Able to give informed consent

Exclusion Criteria:

i. Current cardiopulmonary disease requiring treatment (hypertension permitted) ii. Medical or biophysical conditions that do not permit use of either a cycle ergometer or treadmill iii. MRI contraindications (pacemaker, wires, defibrillator, or implanted heart valves, head surgery requiring aneurysm clips, or any type of electric device (stimulator or pump) implanted in the body) iv. MS exacerbation in the last 30 days v. Pregnant women: Pregnancy status determined by menstrual history and contraceptive method. Confirmatory urine pregnancy test will be used if pregnancy status is uncertain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04 (Actual); Study Completion 2016-05-25 (Actual)

PRIMARY OUTCOMES:
Comparison of correlations in changes in VO2Max at 12 weeks with changes in brain ATP production at 12 weeks between aerobic exercise group and stretching group. | Baseline, Twelve Weeks
  1. Changes in VO2Max testing consists of an aerobic exercise test on a treadmill or stationary bicycle to measure blood pressure, heart rate, and oxygen consumption, and lung function tests
  2. Brain ATP production is measured using a 31P MRSI imaging procedure: MRI data is collected using 7 tesla MRI instrument. All MRI data will be collected within 1.25 hour on each session (2.5 hour total/subject).

SECONDARY OUTCOMES:
Changes in Cognition at 12 weeks | Baseline, Twelve Weeks
  Symbol Digit Modalities Test (SDMT)
Changes in fatigue at 12 weeks | Baseline, Twelve Weeks
  Modified Fatigue Impact Scale (MFIS)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Spain, MD, MSPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States